CLINICAL TRIAL: NCT02686502
Title: Motivation Makes the Move!
Acronym: MoMaMo!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: VTT Technical Research Centre of Finland (Other); Finnish Institute of Occupational Health (Other); University of Western Ontario, Canada (Other); Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Maritta Pöyhönen-Alho, MD, PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TYH2016215; 575/31/2015 (Other Grant/Funding Number: Tekes - the Finnish Funding Agency for Innovation)
Record Dates: First submitted 2016-01-22; First posted 2016-02-19 (Estimated); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Obesity; Cardiovascular Diseases; Physical Conditioning
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Motor Activity | interventions — Exercise; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mode 1 (No Intervention): Current guidelines. Subjects attending the examinations and the tests but not participating the individualized intervention. The subjects will receive general guidance on healthy exercise and diet.
- Mode 2 (Active Comparator): Individualized lifestyle intervention. Exercise intervention will be based on submaximal ergometer test (estimated VO2max), clinical status, personal goals and preferences. Intervention also includes diet counseling, multiprofessional team support, peer support and use of mobile health applications.
  Interventions: Behavioral: Lifestyle
- Mode 3 (Active Comparator): Highly individual lifestyle intervention. In addition to Mode 2 arm intervention optimal intensity zones and volumes for individual exercise training will be determined based on advanced cardiopulmonary exercise test.
  Interventions: Behavioral: Lifestyle

INTERVENTIONS:
Behavioral: Lifestyle — As part of the intervention Mode 2 and 3 subjects will use various mobile health applications including heart rate monitor, global positioning system, diet diary, and weight, sleep and mood monitors. They will also be offered music streaming service for e.g. motivation and relaxation.
  Other Names: Exercise; Diet
  Arms: Mode 2; Mode 3

SUMMARY:
This study evaluates the effect and usability of mobile and cloud technology -based intervention on lifestyle modification in 18-40 year obese and overweight subjects.

The study has a dose-response design with three randomized subjects groups from Mode 1 to Mode 3 with increasing intensity of intervention (guidance, exercise program, diet, support). The special focus of this study is on motivation and use of music and mobile health devices as motivational tools to support individualized exercise training, healthy diet and overall healthy life style.

DETAILED DESCRIPTION:
Obesity negatively impacts health in many ways. It is associated with metabolic diseases and mood disorders and in women pregnancy outcome as well as the health of the offspring.

The modern evolution of societies steers populations towards a profound sedentary lifestyle. Physical activity brings about health benefits, however, the risk reduction for chronic diseases remains significantly greater for fitness than physical activity per se. The recent knowledge suggest Individualized approach rather than general guidelines for exercise in prevention-oriented strategies.

In this study we compare three different intensities of lifestyle intervention: 1) general guidelines for healthy exercise and diet, 2) individual program,and 3) highly individual program. Individual programs will be based on pre-examinations including interview and clinical exercise test. Mobile and cloud technologies will be used to collect data and steer the subjects´ lifestyles and daily activities and together with music to motivate them. The duration of the active intervention is 3 months and it will continue on a self-governing basis up to 1 year. The primary outcome is maximal oxygen consumption (VO2max), and secondary outcomes are physical activity, cardio-respiratory and cardiovascular parameters, blood volume, total hemoglobin mass, metabolic health along with chronic low-grade inflammation and well-being.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 27,5 kg/m2
* estimated by health care personnel to benefit from lifestyle modification

Exclusion Criteria:

* inability to perform exercise testing and intervention (physical, mental or other reason)
* not able to operate in Finnish (some applications only in Finnish for the time being)
* severe anemia (Hb<108 g/l for women and < 124 g/l for men)
* smoking (disturbs autonomic nervous system measurements)
* regular medication affecting glucose metabolism (excluding insulin) or autonomic nervous system (e.g. beta blockers, SSRI)
* ongoing pregnancy or breast feeding
* prisoner

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-04; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change from measured baseline maximal O2 uptake (VO2max) at 3 months | 3 months

SECONDARY OUTCOMES:
Change from baseline quality of life at 3 months | 3 months
  Rand-36 questionnaire
Change from baseline total plasma cholesterol at 3 months | 3 months
Change from baseline physical activity at 3 months | 3 months
  The International Physical Activity Questionnaire short version (IPAQ-S)
Change from baseline body weight at 3 months | 3 months
  weight in kilograms
Change from baseline quality of life at 1 year | 1 year
  Rand-36 questionnaire
Change from baseline physical activity at 1 year | 1 year
  The International Physical Activity Questionnaire short version (IPAQ-S)
Change from baseline body weight at 1 year | 1 year
  weight in kilograms
Change from baseline total plasma cholesterol at 1 year | 1 year
Change from baseline plasma HDL cholesterol at 3 months | 3 months
Change from baseline plasma HDL cholesterol at 1 year | 1 year
Change from baseline plasma LDL cholesterol at 3 months | 3 months
Change from baseline plasma LDL cholesterol at 1 year | 1 year
Change from baseline plasma triglycerides at 3 months | 3 months
Change from baseline plasma triglycerides at 1 year | 1 year
Change from baseline blood glucose balance at 3 months | 3 months
  Blood glucose balance assessed by 75-g 2 h oral glucose tolerance test
Change from baseline blood glucose balance at 1 year | 1 year
  Blood glucose balance assessed by 75-g 2 h oral glucose tolerance test
Change from baseline fasting plasma insulin at 3 months | 3 months
Change from baseline fasting plasma insulin at 1 year | 1 year
Change from baseline body composition at 3 months | 3 months
  Body composition assessed by bioimpedance
Change from baseline mood at 3 months | 3 months
  PANAS questionnaire
Change from baseline mood at 1 year | 1 year
  PANAS questionnaire
Change from baseline work productivity at 3 months | 3 months
  Work Productivity and Activity Impairment Questionnaire (WPAI)
Change from baseline work productivity at 1 year | 1 year
  Work Productivity and Activity Impairment Questionnaire (WPAI)
Change from baseline sexual functions at 3 months (females) | 3 months
  The Female Sexual Function Index (FSFI)
Change from baseline sexual functions at 1 year (females) | 1 year
  The Female Sexual Function Index (FSFI)
Change from baseline music consumption at 3 months | 3 months
  Music in Mood Regulation questionnaire (MMR)
Change from baseline music consumption at 1 year | 1 year
  Music in Mood Regulation questionnaire (MMR)
Change from baseline calorie intake at 3 months | 3 months
  Food diary filled during 3 consecutive days every 2 weeks
Change from baseline calorie intake at 1 year | 1 year
  Food diary filled during 3 consecutive days every 2 weeks
Change from baseline heart rate variability at 3 months | 3 months
  3 day electrocardiography monitoring
Change from baseline heart rate variability at 1 year | 1 year
  3 day electrocardiography monitoring
Change from baseline protein intake at 3 months | 3 months
  Food diary filled during 3 consecutive days every 2 weeks
Change from baseline protein intake at 1 year | 1 year
  Food diary filled during 3 consecutive days every 2 weeks
Change from baseline fat intake at 3 months | 3 months
  Food diary filled during 3 consecutive days every 2 weeks
Change from baseline fat intake at 1 year | 1 year
  Food diary filled during 3 consecutive days every 2 weeks
Change from baseline carbohydrate intake at 3 months | 3 months
  Food diary filled during 3 consecutive days every 2 weeks
Change from baseline carbohydrate intake at 1 year | 1 year
  Food diary filled during 3 consecutive days every 2 weeks
Height | 0 months
  height measured in centimeters
Stability of personality | 0 months
  Five Factor Personality test
Stability of personality | 3 months
  Five Factor Personality test
Stability of personality | 1 year
  Five Factor Personality test
Change from baseline depression at 3 months | 3 months
  Beck questionnaire
Change from baseline depression at 1 year | 1 year
  Beck questionnaire
Change from baseline waist-hip-ratio at 3 months | 3 months
Change from baseline waist-hip-ratio at 1 year | 1 year
Change from baseline plasma ferritin (P-Ferrit) level at 3 months | 3 months
Change from baseline plasma ferritin (P-Ferrit) level at 1 year | 1 year
Change from baseline plasma transferrin receptor (P-TfR) level at 3 months | 3 months
Change from baseline plasma transferrin receptor (P-TfR) level at 1 year | 1 year
Change from baseline plasma sensitive C-reactive protein (CRP) level at 3 months | 3 months
Change from baseline plasma sensitive C-reactive protein (CRP) level at 1 year | 1 year
Change from baseline plasma tumor necrosis factor alpha alpha (P-TNF alpha) level at 3 months | 3 months
Change from baseline plasma tumor necrosis factor alpha alpha (P-TNF alpha) level at 1 year | 1 year
Change from baseline plasma Interleukin-6 (IL6) level at 3 months | 3 months
Change from baseline plasma Interleukin-6 (IL-6) level at 1 year | 1 year
Change from baseline plasma Interleukin-10 (IL-10) level at 3 months | 3 months
Change from baseline plasma IInterleukin-10 (IL-10) level at 1 year | 1 year
Change from baseline plasma Interleukin-15 (IL-15) level at 3 months | 3 months
Change from baseline plasma Interleukin-15 (IL-15) level at 1 year | 1 year
Change from baseline plasma Interleukin-8 (IL-8) level at 3 months | 3 months
Change from baseline plasma Interleukin-8 (IL-8) level at 1 year | 1 year
Change from baseline plasma Interleukin-1 beta (IL-1 beta) level at 3 months | 3 months
Change from baseline plasma Interleukin-1 beta (IL-1 beta) level at 1 year | 1 year
Change from baseline body mass index (BMI) at 3 months | 3 months
  BMI in kg/m^2
Change from baseline body mass index (BMI) at 1 year | 1 year
  BMI in kg/m^2
Change from estimated (non-exercise questionnaire) baseline maximal O2 uptake (VO2max) at 3 months | 3 months
Change from estimated (non-exercise questionnaire) baseline maximal O2 uptake (VO2max) at 1 year | 1 year
Change from estimated (step test) baseline VO2max at 3 months | 3 months
Change from estimated (step test) baseline VO2max at 1 year | 1 year
Change from estimated (submaximal cycle ergometer exercise) baseline VO2max at 3 months | 3 months
Change from baseline maximal work rate (WR) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) pulmonary ventilation (VE) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) alveolar ventilation (VA) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) breathing frequency (Bf) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) tidal volume (VT) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) tidal volume - dead space ratio (VD/VT) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) end tidal O2 (PETO2) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) end tidal CO2 (PETCO2) at 3 months | 3 months
Change from baseline submaximal (work rate specific) VO2 at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) CO2 production (VCO2) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) respiratory exchange ratio (RER) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) ventilatory equivalent for O2 uptake (VE/VO2) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) ventilatory equivalent for CO2 production (VE/VCO2) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) O2 pulse (VO2/HR) at 3 months | 3 months
Change from baseline resting heart rate (HR) at 3 months | 3 months
Change from baseline resting heart rate (HR) at 1 year | 1 year
Change from baseline resting blood pressure (BP, systolic, diastolic, pulse, mean) at 3 months | 3 months
Change from baseline resting blood pressure (BP, systolic, diastolic, pulse, mean) at 1 year | 1 year
Change from baseline maximal and submaximal (work rate specific) heart rate (HR) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) arterial blood pressure (BP, systolic, diastolic, pulse, mean) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) cardiac output (Q) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) stroke volume (SV) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) end-diastolic volume (EDV) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) ejection fraction (EF) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) cardiac index at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) contractility index at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) estimate of left ventricular ejection time at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) left cardiac work index at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) early diastolic function ratio at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) calculated arteriovenous O2 difference ((a-v)O2) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) arterial O2 saturation (SpO2) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) calculated arterial O2 content (CaO2) heart rate (HR) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) calculated O2 delivery (QaO2) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) calculated O2 extraction (O2ext) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) calculated systemic vascular resistance (SVR) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) metabolic equivalent (MET) at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) tissue saturation index (TSI) in skeletal muscle and cerebral tissue at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) oxyhemoglobin concentration (O2Hb) in skeletal muscle and cerebral tissue at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) deoxyhemoglobin concentration (HHb) in skeletal muscle and cerebral tissue at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) total hemoglobin concentration (Hbtot) in skeletal muscle and cerebral tissue at 3 months | 3 months
Change from baseline maximal and submaximal (work rate specific) estimated regional blood flow (BFe) at 3 months | 3 months
Change from baseline ankle-brachial blood pressure index (ABI) at 3 months | 3 months
Change from baseline cardio-ankle vascular index (CAVI) at 3 months | 3 months
Change from baseline blood pressure variability (BPV) at 3 months | 3 months
Change from baseline baroreflex sensitivity (BRS) at 3 months | 3 months
Change from baseline postural sway during orthostatic test at 3 months | 3 months
Change from baseline nocturnal heart rate variability (HRVn) at 3 months | 3 months
Change from baseline heart rate on-kinetics and off-kinetics during an exercise test at 3 months | 3 months
Change from baseline alveolar gas exchange on-kinetics and off-kinetics during an exercise test at 3 months | 3 months
Change from baseline tissue oxygenation on-kinetics and off-kinetics during an exercise test at 3 months | 3 months
Change from baseline hemoglobin concentration ([Hb]) at 3 months | 3 months
Change from baseline hemoglobin concentration ([Hb]) at 1 year | 1 year
Change from baseline hematocrit (Hct) at 3 months | 3 months
Change from baseline hematocrit (Hct) at 1 year | 1 year
Change from baseline blood count at 3 months | 3 months
Change from baseline blood count at 1 year | 1 year
Change from baseline blood volume (BV) at 3 months | 3 months
Change from baseline total hemoglobin mass (tHb-mass]) at 3 months | 3 months
Change from baseline erythrocyte volume (EV) at 3 months | 3 months
Change from baseline erythrocyte volume (EV) at 1 year | 1 year
Change from baseline plasma volume (PV) at 3 months | 3 months
Change from baseline glycosylated hemoglobin (HbA1c) at 3 months | 3 months
Change from baseline glycosylated hemoglobin (HbA1c) at 1 year | 1 year
Change from baseline homeostasis model assessment of insulin resistance (HOMA-IR) at 3 months | 3 months
Change from baseline homeostasis model assessment of insulin resistance (HOMA-IR) at 1 year | 1 year
Change from baseline blood interleukin 2 (IL-2) at 3 months | 3 months
Change from baseline blood interleukin 2 (IL-2) at 1 year | 1 year
Change from baseline blood interleukin (IL-4) at 3 months | 3 months
Change from baseline blood interleukin (IL-4) at 1 year | 1 year
Change from baseline blood interleukin 5 (IL-5) at 3 months | 3 months
Change from baseline blood interleukin 5 (IL-5) at 1 year | 1 year
Change from baseline blood granulocyte-macrophage colony-stimulating factor (GM-CSF) at 3 months | 3 months
Change from baseline blood granulocyte-macrophage colony-stimulating factor (GM-CSF) at 1 year | 1 year
Change from baseline blood interferon gamma (IFNγ) at 3 months | 3 months
Change from baseline blood interferon gamma (IFNγ) at 1 year | 1 year
Change from baseline blood resistin at 3 months | 3 months
Change from baseline blood resistin at 1 year | 1 year
Change from baseline blood leptin at 3 months | 3 months
Change from baseline blood leptin at 1 year | 1 year
Change from baseline blood adiponectin at 3 months | 3 months
Change from baseline blood adiponectin at 1 year | 1 year
Change from baseline Forced Vital Capacity (FVC) at 3 months | 3 months
Change from baseline Forced Expiratory Volume in the 1st second (FEV1) at 3 months | 3 months
Change from baseline The percentage of total expired volume that was expired in the first second (FEV1%) at 3 months | 3 months
Change from baseline Forced Inspiratory Vital Capacity (FIV) at 3 months | 3 months
Change from baseline Peak Expiratory Flow (PEF) at 3 months | 3 months
Change from baseline Peak Inspiratory Flow (PIF) at 3 months | 3 months
Change from baseline Forced Expiratory Flow between 25% and 75% of FVC (FEF2575) at 3 months | 3 months
Change from baseline Forced Expiratory Flow at 25% of expired volume during FVC test (FEF25) at 3 months | 3 months
Change from baseline Forced Expiratory Flow at 50% of expired volume during FVC test (FEF50) at 3 months | 3 months
Change from baseline Forced Expiratory Flow at 75% of expired volume during FVC test (FEF75) at 3 months | 3 months
Change from baseline Forced Expiratory Time (FET) at 3 months | 3 months
Change from baseline sleep time cumulatively to 3 months | 3 months
Change from baseline sleep time cumulatively to 1 year | 1 year
Change from baseline self-reported feelings on him-/herself, health, outlook, intimate relationship/marriage, family, friends, sex, work, studies, hobbies, money, pets, technology and traffic cumulatively to 3 months | 3 months
Change from baseline self-reported feelings on him-/herself, health, outlook, intimate relationship/marriage, family, friends, sex, work, studies, hobbies, money, pets, technology and traffic cumulatively to 1 year | 1 year
Change from baseline possible obstructive sleep apnea (OSA) to 3 months | 3 months
Change from baseline calculated Wellness Index (WI) at 3 months | 3 months
Change from baseline calculated Wellness Index (WI) at 1 year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Seppo Heinonen, Professor, Study Director — HUCH, Dept. of Obstetrics and Gynecology
Locations (2):
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Vantaa Health Care and Social Services, Vantaa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaseva K, Tervaniemi M, Heikura E, Kostilainen K, Poyhonen-Alho M, Shoemaker JK, Petrella RJ, Peltonen JE. Identifying Personality Characteristics and Indicators of Psychological Well-Being Associated With Attrition in the Motivation Makes the Move! Physical Activity Intervention: Randomized Technology-Supported Trial. JMIR Form Res. 2022 Nov 25;6(11):e30285. doi: 10.2196/30285. PMID 36427239